CLINICAL TRIAL: NCT06509958
Title: A Phase Ⅱ Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Single Injection Adductor Canal Block With HR18034 for Postoperative Pain Management in Total Knee Arthroplasty
Brief Title: Phase Ⅱ Study of Adductor Canal Block With HR18034 for Postsurgical Pain Management in TKA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's R&D Strategy adjusted
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR18034-204
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain Management in Total Knee Arthroplasty
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental)
  Interventions: Drug: HR18034
- Dose 2 (Experimental)
  Interventions: Drug: HR18034
- Ropivacaine Hydrochloride Injection (Active Comparator)
  Interventions: Drug: Ropivacaine Hydrochloride Injection

INTERVENTIONS:
Drug: HR18034 — HR18034
  Arms: Dose 1; Dose 2
Drug: Ropivacaine Hydrochloride Injection — Ropivacaine Hydrochloride Injection
  Arms: Ropivacaine Hydrochloride Injection

SUMMARY:
Phase Ⅱ, randomized, double-blind, comparator-controlled study to evaluate the efficacy, safety and pharmacokinetics of single injection adductor canal block with HR18034 for postoperative pain management in total knee arthroplasty compared with ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Scheduled to undergo primary unilateral total knee arthroplasty under general anesthesia.
3. Male or female，aged ≥ 18 years
4. Body mass index (BMI) ≥ 18 kg/m2
5. American Society of Anesthesiologists (ASA) Physical Status Classification Ⅰ~Ⅲ

Exclusion Criteria:

1. Subjects with deformity of the involving operative limb, or other neuropathy
2. Subjects with a history of new myocardial infarction or unstable angina within 6 months prior to randomization;
3. Subjects with a history of ischemic stroke or transient ischemic attack (TIA)
4. Subjects with a history of mental system diseases and cognitive dysfunction
5. Combination of other pain conditions that may affect postoperative pain assessment
6. Persistent or recurrent nausea and/or vomiting due to other etiologies, including, but not limited to gastric outlet obstruction, hypercalcemia, or active peptic ulcer
7. Subjects with a history of deep vein thrombosis-related disease
8. Clinically significant abnormal clinical laboratory test value
9. Allergic to a drug ingredient or component
10. Use of any of medications, which affect drug metabolism or analgesia evaluation, within 5 half-lives or as specified prior to the study surgical procedure
11. History of alcohol abuse or prescription and/or illicit drug abuse
12. Pregnant or nursing women
13. No birth control during the specified period of time
14. Participated in clinical trials of other drugs (received experimental drugs)
15. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
AUC0-72h of the NRS-A pain intensity scores. | 0 to 72 hours
  AUC of NRS pain intensity scores at activity (NRS-A) through 72 hours after the beginning of study drug administration.

SECONDARY OUTCOMES:
AUC of the NRS-A pain intensity scores. | 0-24, 0-48hours
  AUC of NRS pain intensity scores at activity (NRS-A) for time periods 0-24, 0-48 hours.
AUC of the NRS-R pain intensity scores. | 0-24, 0-48，0-72 hours
AUC of NRS pain intensity scores at rest (NRS-R) for time periods 0-24, 0-48 ,0-72 hours. | 0-24, 0-48 ,0-72 hours.
Pain intensity assessed using an 12-point NRS ranging. | Baseline till 72 hours after the beginning of study drug administration
Proportion of subjects who used no rescue opioid analgesic. | 0-24, 24-48, 48-72, 0-72 hours
Total rescue analgesic consumption. | 0-24, 24-48, 48-72, 0-72 hours
Time to the first postoperative use of rescue opioid analgesics. | 0-72hours
Quadriceps muscle strength score. | Baseline till 72 hours after the beginning of study drug administration
Range of motion of the knee joint. | Baseline till 72 hours after the beginning of study drug administration
Subjects' satisfaction rating | 72 hours
Investigators' satisfaction rating | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided